CLINICAL TRIAL: NCT05573321
Title: Effect of Blood Flow Restriction Exercise on Acute Systemic Irisin, Myostatin and Decorin Levels
Brief Title: The Effect of Blood Flow Restriction (Bfr) Exercise on Acute Systemic Myokine Levels in Healthy Trained Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Goksu Gokce, Sports Medicine Resident, Ege University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 22-7T/59
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Muscle Hypotrophy
Keywords: blood flow restriction; myokines
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR-RE (Experimental): In the BFR-RE intervention, the exercise will be done as a set of 30 repetitions with a loading of 30% of 1 RM and an additional 3 sets x 15 repetitions, with 30 seconds rest between sets.
  Interventions: Other: BFR-RE; Other: HL-RE
- HL-RE (Active Comparator): In the HL-RE intervention, the exercise will be performed with a loading of 80% of 1 RM, with 4 sets x 7 repetitions, with 60 seconds of rest between sets.
  Interventions: Other: BFR-RE; Other: HL-RE

INTERVENTIONS:
Other: BFR-RE — In the BFR-RE intervention, the exercise will be done as a set of 30 repetitions with a loading of 30% of 1 RM and an additional 3 sets x 15 repetitions, with 30 seconds rest between sets. In both groups, bilateral leg extension exercise will be performed by using the leg extension machine for resistance exercise. In the blood flow restriction group (BFR-RE), the cuff will be placed in the proximal region of the thigh bilaterally, inflated to a pressure equivalent to 50% of the estimated arterial occlusion pressure (AOP), and leg extension exercise will be performed under this condition. In the BFR-RE group, the blood flow restriction time will be between 5-10 minutes. Venous blood samples will be collected from the arm antecubital region of the participants just before the exercise session, immediately after the exercise, and 1 hour after the exercise. Plasma irisin, myostatin and decorin levels will be measured from the samples taken.
Other: HL-RE — In the HL-RE intervention, the exercise will be performed with a loading of 80% of 1 RM, with 4 sets x 7 repetitions, with 60 seconds of rest between sets. In both groups, bilateral leg extension exercise will be performed by using the leg extension machine for resistance exercise. Venous blood samples will be collected from the arm antecubital region of the participants just before the exercise session, immediately after the exercise, and 1 hour after the exercise. Plasma irisin, myostatin and decorin levels will be measured from the samples taken.

SUMMARY:
The aim of the study is to measure and compare acute systemic irisin, myostatin and decorin levels after a single session of blood flow restricted resistance exercise and resistance exercise without blood flow restriction in healthy, trained male participants aged 18-35 years. For this purpose, a total of 22 people will be included in the study. Participants will be randomly allocated to 2 exercise groups as resistance exercise with blood flow restriction (BFR-RE) and resistance exercise without blood flow restriction (HL-RE) and will be subjected to cross-over. In the HL-RE intervention, the exercise will be performed with a loading of 80% of 1 RM, with 4 sets x 7 repetitions, with 60 seconds of rest between sets. In the BFR-RE intervention, the exercise will be done as a set of 30 repetitions with a loading of 30% of 1 RM and an additional 3 sets x 15 repetitions, with 30 seconds rest between sets. Total exercise volumes were tried to be equalized and skeletal muscle hypertrophy was selected in accordance with exercise guidelines. In both groups, bilateral leg extension exercise will be performed using the leg extension machine for resistance exercise. In the blood flow restriction group (BFR-RE), the cuff will be placed in the proximal region of the thigh bilaterally, inflated to a pressure equivalent to 50% of the estimated arterial occlusion pressure (AOP), and leg extension exercise will be performed under this condition. In the BFR-RE group, the blood flow restriction time will be between 5-10 minutes. Exercise sessions will be conducted under supervision. Venous blood samples will be collected from the arm antecubital region of the participants just before the exercise session, immediately after the exercise, and 1 hour after the exercise. Plasma irisin, myostatin and decorin levels will be measured from the samples taken. It is well known that resistance exercise is important in maintaining and increasing muscle mass (hypertrophy). Studies have shown the involvement of certain myokines in skeletal muscle hypertrophy, although few studies have been conducted on the systemic response of myokines to BFR-RE that may play a potential role in hypertrophy. Therefore, the planned study aimed to reveal the similarities or differences in the systemic myokine response between BFR-RE and HL-RE.

DETAILED DESCRIPTION:
Resistance exercise is a type of exercise classically used to increase skeletal muscle hypertrophy and muscle strength. Resistance training is an important component of training in most sports, and it also plays a role in injury prevention and rehabilitation. In dynamic resistance exercise, the intensity is usually determined by measuring the maximum weight that can be lifted only once (one repetition maximum, 1RM). The American College of Sports Medicine (ACSM) recommends more than 70% of 1RM to increase muscle mass (high load resistance exercise, HL-RE). High-intensity loads recommended by the ACSM may not be a suitable option for populations with sarcopenia, the elderly with chronic health conditions, or those with injuries that cannot tolerate heavy load, as they create excessive mechanical stress on the tissues during exercise and pose a potential risk of injury. There is increasing evidence that the use of blood flow restriction (BFR), also known as occlusion or Kaatsu training, with low-load resistance exercise (<50% 1RM) provides hypertrophic gains. This training method (BFR RE) is an exercise method performed by placing an inflatable cuff on the proximal part of the extremity (arm or leg) to restrict blood flow and restricting venous return distal to the obstruction without obstructing arterial flow. As publications using this method increase, interest in BFR-RE has increased to increase skeletal muscle hypertrophy and strength in athletes, the elderly, or clinical populations (such as cerebrovascular, cardiac, neuromuscular diseases, obesity). Standard hypertrophy exercise parameters consist of 1-3 total sets, 8-12 repetitions for sets, and 1-2 minutes rest between sets, with a loading of 70-85% of 1RM in beginner-intermediate levels. BFR-RE, on the other hand, consists of a loading interval of 20-40% of 1RM, a set of 30 repetitions, followed by 3 additional sets of 15 repetitions, with 30 seconds of rest between sets. Despite this difference in exercise protocols, both approaches provide skeletal muscle hypertrophy. Studies show that low-load-high-rep resistance exercises, when performed until fatigue, cause skeletal muscle hypertrophy similar to high-load-low-rep resistance exercises. In addition, BFR-RE is superior to unrestricted low-load resistance exercise in terms of skeletal muscle hypertrophy when the exercise volume is equalized. According to a meta-analysis, BFR-RE has been shown to induce increases in muscle mass comparable to HL-RE regardless of absolute occlusion pressure, cuff width, and method of generating occlusion pressure. Although the potent hypertrophic effects of BFR-RE have been demonstrated by numerous studies, the underlying mechanisms responsible for such effects are not well defined. Although the potent hypertrophic effects of BFR-RE have been demonstrated by numerous studies, the underlying mechanisms responsible for such effects are not well defined. Metabolic stress (accumulation of metabolites as a result of the ischemic/hypoxic environment) has been suggested to be the primary responsible factor, and is thought to activate numerous other mechanisms thought to induce muscle hypertrophy through autocrine and/or paracrine actions. Secondary mechanisms activated by metabolic stress include involvement of fast twitch muscle fibers (type 2 fibers), release of certain hormones (GH, IGF-1), myokine production, production of reactive oxygen products and cell swelling. However, it is important to recognize that some of these mechanisms are largely induced not by metabolic stress but rather by mechanical tension (another primary factor of muscle hypertrophy). Given that mechanical strain is typically low (<50% 1RM) in BFR-RE, the extent of its involvement in hypertrophic adaptations is questionable. However, mechanical tension and metabolic stress, which are ultimately the primary factors responsible for hypertrophy, act synergistically to produce muscle hypertrophy in BFR-RE. Cytokines are a large family of polypeptides and proteins that function as intercellular messengers. While their primary function is typically associated with immune response, many cytokines appear to exhibit functional pleiotropy. A cytokine may mediate different effects depending on the initial stimulus, the target cell, or other co-released cytokines. Cytokines can also act locally (autocrine or paracrine) or systemically (endocrine) depending on the target tissue. Skeletal muscle has been found to release cytokines in response to muscle contraction. These cytokines, called myokines, have local effects on muscle as well as systemic effects on other tissues. Myokine release after muscle contraction varies according to the intensity, mode and volume of the exercise performed by the person. There are theories that metabolic stress may mediate muscle hypertrophy by upregulating anabolic myokines and/or downregulating catabolic myokines. Irisin was discovered by Bostrom et al in 2012 as a PGC-1α (peroxisome proliferator-activated receptor coactivator 1-alpha)-dependent myokine. It is proteolytically cleaved from the membrane protein FDNC-5 (fibronectin domain-containing protein-5) and secreted from skeletal muscle into the circulation in response to exercise. Irisin is a myokine primarily known for its effect on the conversion of white adipose tissue to brown adipose tissue, thereby increasing thermogenesis and energy metabolism. However, there is new evidence suggesting that the iris may have a role in regulating muscle hypertrophy. Recent studies show that acute intense resistance exercise increases circulating irisin concentrations. It has been reported that irisin induces skeletal muscle hypertrophy and reduces denervation-induced atrophy by activating IL-6 in rodents. It also suggests that irisin may play a role in skeletal muscle hypertrophy by upregulating IGF-1 and downregulating myostatin in human myocyte cultures and in vitro treatment with irisin. Myostatin is a member of the TGF-ß (transforming growth factor-beta) family and acts as a negative regulator of skeletal muscle development. High myostatin levels are significantly associated with muscle wasting diseases, myopathy and sarcopenia. A significant increase in muscle mass was observed in individuals with mutations in both copies of the myostatin gene compared to normal individuals. There are studies showing that myostatin level decreases with a single session of resistance exercise. It has been shown that myostatin levels in the plantaris muscle of rats following blood flow restricted exercise (BFR) were significantly reduced compared to the sham group. Decorin has been defined as another myokine that plays a role in muscle hypertrophy. Myotubes secrete decorin and decorin regulates protein synthesis in vitro. In addition, in vivo evidence from rodent skeletal muscle has shown that overexpression of decorin can upregulate several factors involved in inhibiting myostatin, a potent myokine that decreases muscle cell growth and differentiation and increases protein degradation. It is believed that decorin may be involved in anabolic activity in skeletal muscle by inhibiting myostatin. It has been shown that various acute resistance exercises (LL-RE, HL-RE, BFR-RE) result in a systemic release of decorin, and this myokine may be involved in the hypertrophic response to resistance exercise. There appears to be a lack of research investigating the potential role played by myokines in BFR-RE-induced skeletal muscle hypertrophy. The aim of this study is to evaluate the systemic irisin, myostatin and decorin myokines levels after acute BFR-RE and HL-RE, and to measure whether BFR-RE alters the exercise-induced myokine response. We predict that systemic irisin, myostatin and decorin myokine responses to BFR-RE and HL-RE will be similar.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18-35 years old and male gender
2. To have been doing resistance exercises for at least 1 year and to be accustomed to lower extremity resistance exercises
3. Not doing any resistance exercise with restricted blood flow in the last 1 month
4. Not doing lower extremity resistance exercise for at least 48 hours
5. Answering no to all questions in the Exercise Readiness Questionnaire (EGZ-A+)

Exclusion Criteria:

1. Presence of musculoskeletal injury or disability that may prevent exercise with restricted blood flow
2. Using non-steroidal anti-inflammatory drugs (NSAIDs) or supplements that may have an anti-inflammatory effect
3. Being at risk for cardiovascular disease
4. Regular use of tobacco products
5. Using ergogenic support

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-02-14 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
change in irisin concentrations | immediately before the exercise session, immediately after the exercise and 1 hour after the exercise
  It was discovered by Bostrom et al in 2012 as a PGC-1α (peroxisome proliferator-activated receptor coactivator 1-alpha)-dependent myokine. It is proteolytically cleaved from the membrane protein FDNC-5 (fibronectin domain containing protein-5) and secreted from skeletal muscle into the circulation in response to exercise. Irisin is a myokine mainly known for its effect on the conversion of white adipose tissue to brown adipose tissue, thereby increasing thermogenesis and energy metabolism. However, there is new evidence to suggest that the iris may have a role in regulating muscle hypertrophy.
change in myostatin concentrations | immediately before the exercise session, immediately after the exercise and 1 hour after the exercise
  It is a member of the TGF-ß (transforming growth factor-beta) family and acts as a negative regulator of skeletal muscle growth.
change in decorin concentrations | immediately before the exercise session, immediately after the exercise and 1 hour after the exercise
  It has been identified as another myokine that plays a role in muscle hypertrophy. Decorin is thought to be involved in anabolic activity in skeletal muscle by inhibiting myostatin.

CONTACTS AND LOCATIONS:
Overall Officials: Metin Ergun, Study Chair — Ege University Hospital, Sports Medicine Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Background] Yasuda T, Ogasawara R, Sakamaki M, Bemben MG, Abe T. Relationship between limb and trunk muscle hypertrophy following high-intensity resistance training and blood flow-restricted low-intensity resistance training. Clin Physiol Funct Imaging. 2011 Sep;31(5):347-51. doi: 10.1111/j.1475-097X.2011.01022.x. Epub 2011 Mar 22. PMID 21771252
- [Background] Pope ZK, Willardson JM, Schoenfeld BJ. Exercise and blood flow restriction. J Strength Cond Res. 2013 Oct;27(10):2914-26. doi: 10.1519/JSC.0b013e3182874721. PMID 23364292
- [Background] Wilk M, Krzysztofik M, Gepfert M, Poprzecki S, Golas A, Maszczyk A. Technical and Training Related Aspects of Resistance Training Using Blood Flow Restriction in Competitive Sport - A Review. J Hum Kinet. 2018 Dec 31;65:249-260. doi: 10.2478/hukin-2018-0101. eCollection 2018 Dec. PMID 30687436
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Background] Martin-Hernandez J, Marin PJ, Menendez H, Ferrero C, Loenneke JP, Herrero AJ. Muscular adaptations after two different volumes of blood flow-restricted training. Scand J Med Sci Sports. 2013 Mar;23(2):e114-20. doi: 10.1111/sms.12036. Epub 2012 Dec 27. PMID 23278841
- [Background] Slysz J, Stultz J, Burr JF. The efficacy of blood flow restricted exercise: A systematic review & meta-analysis. J Sci Med Sport. 2016 Aug;19(8):669-75. doi: 10.1016/j.jsams.2015.09.005. Epub 2015 Sep 28. PMID 26463594
- [Background] Mitchell CJ, Churchward-Venne TA, West DW, Burd NA, Breen L, Baker SK, Phillips SM. Resistance exercise load does not determine training-mediated hypertrophic gains in young men. J Appl Physiol (1985). 2012 Jul;113(1):71-7. doi: 10.1152/japplphysiol.00307.2012. Epub 2012 Apr 19. PMID 22518835
- [Background] Morton RW, Oikawa SY, Wavell CG, Mazara N, McGlory C, Quadrilatero J, Baechler BL, Baker SK, Phillips SM. Neither load nor systemic hormones determine resistance training-mediated hypertrophy or strength gains in resistance-trained young men. J Appl Physiol (1985). 2016 Jul 1;121(1):129-38. doi: 10.1152/japplphysiol.00154.2016. Epub 2016 May 12. PMID 27174923
- [Background] Takarada Y, Tsuruta T, Ishii N. Cooperative effects of exercise and occlusive stimuli on muscular function in low-intensity resistance exercise with moderate vascular occlusion. Jpn J Physiol. 2004 Dec;54(6):585-92. doi: 10.2170/jjphysiol.54.585. PMID 15760491
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Background] Lixandrao ME, Ugrinowitsch C, Berton R, Vechin FC, Conceicao MS, Damas F, Libardi CA, Roschel H. Magnitude of Muscle Strength and Mass Adaptations Between High-Load Resistance Training Versus Low-Load Resistance Training Associated with Blood-Flow Restriction: A Systematic Review and Meta-Analysis. Sports Med. 2018 Feb;48(2):361-378. doi: 10.1007/s40279-017-0795-y. PMID 29043659
- [Background] Loenneke JP, Fahs CA, Wilson JM, Bemben MG. Blood flow restriction: the metabolite/volume threshold theory. Med Hypotheses. 2011 Nov;77(5):748-52. doi: 10.1016/j.mehy.2011.07.029. Epub 2011 Aug 12. PMID 21840132
- [Background] Moritani T, Sherman WM, Shibata M, Matsumoto T, Shinohara M. Oxygen availability and motor unit activity in humans. Eur J Appl Physiol Occup Physiol. 1992;64(6):552-6. doi: 10.1007/BF00843767. PMID 1618195
- [Background] Yasuda T, Brechue WF, Fujita T, Shirakawa J, Sato Y, Abe T. Muscle activation during low-intensity muscle contractions with restricted blood flow. J Sports Sci. 2009 Mar;27(5):479-89. doi: 10.1080/02640410802626567. PMID 19253083
- [Background] Takarada Y, Nakamura Y, Aruga S, Onda T, Miyazaki S, Ishii N. Rapid increase in plasma growth hormone after low-intensity resistance exercise with vascular occlusion. J Appl Physiol (1985). 2000 Jan;88(1):61-5. doi: 10.1152/jappl.2000.88.1.61. PMID 10642363
- [Background] Reeves GV, Kraemer RR, Hollander DB, Clavier J, Thomas C, Francois M, Castracane VD. Comparison of hormone responses following light resistance exercise with partial vascular occlusion and moderately difficult resistance exercise without occlusion. J Appl Physiol (1985). 2006 Dec;101(6):1616-22. doi: 10.1152/japplphysiol.00440.2006. Epub 2006 Aug 10. PMID 16902061
- [Background] Kaijser L, Sundberg CJ, Eiken O, Nygren A, Esbjornsson M, Sylven C, Jansson E. Muscle oxidative capacity and work performance after training under local leg ischemia. J Appl Physiol (1985). 1990 Aug;69(2):785-7. doi: 10.1152/jappl.1990.69.2.785. PMID 2146245
- [Background] Loenneke JP, Fahs CA, Rossow LM, Abe T, Bemben MG. The anabolic benefits of venous blood flow restriction training may be induced by muscle cell swelling. Med Hypotheses. 2012 Jan;78(1):151-4. doi: 10.1016/j.mehy.2011.10.014. Epub 2011 Nov 1. PMID 22051111
- [Background] Peake JM, Della Gatta P, Suzuki K, Nieman DC. Cytokine expression and secretion by skeletal muscle cells: regulatory mechanisms and exercise effects. Exerc Immunol Rev. 2015;21:8-25. PMID 25826432
- [Background] Bostrom P, Wu J, Jedrychowski MP, Korde A, Ye L, Lo JC, Rasbach KA, Bostrom EA, Choi JH, Long JZ, Kajimura S, Zingaretti MC, Vind BF, Tu H, Cinti S, Hojlund K, Gygi SP, Spiegelman BM. A PGC1-alpha-dependent myokine that drives brown-fat-like development of white fat and thermogenesis. Nature. 2012 Jan 11;481(7382):463-8. doi: 10.1038/nature10777. PMID 22237023
- [Background] Huh JY, Dincer F, Mesfum E, Mantzoros CS. Irisin stimulates muscle growth-related genes and regulates adipocyte differentiation and metabolism in humans. Int J Obes (Lond). 2014 Dec;38(12):1538-44. doi: 10.1038/ijo.2014.42. Epub 2014 Mar 11. PMID 24614098
- [Background] Nygaard H, Slettalokken G, Vegge G, Hollan I, Whist JE, Strand T, Ronnestad BR, Ellefsen S. Irisin in blood increases transiently after single sessions of intense endurance exercise and heavy strength training. PLoS One. 2015 Mar 17;10(3):e0121367. doi: 10.1371/journal.pone.0121367. eCollection 2015. PMID 25781950
- [Background] Tsuchiya Y, Ando D, Takamatsu K, Goto K. Resistance exercise induces a greater irisin response than endurance exercise. Metabolism. 2015 Sep;64(9):1042-50. doi: 10.1016/j.metabol.2015.05.010. Epub 2015 May 29. PMID 26081427
- [Background] Reza MM, Subramaniyam N, Sim CM, Ge X, Sathiakumar D, McFarlane C, Sharma M, Kambadur R. Irisin is a pro-myogenic factor that induces skeletal muscle hypertrophy and rescues denervation-induced atrophy. Nat Commun. 2017 Oct 24;8(1):1104. doi: 10.1038/s41467-017-01131-0. PMID 29062100
- [Background] Roth SM, Walsh S. Myostatin: a therapeutic target for skeletal muscle wasting. Curr Opin Clin Nutr Metab Care. 2004 May;7(3):259-63. doi: 10.1097/00075197-200405000-00004. PMID 15075916
- [Background] Gonzalez-Cadavid NF, Taylor WE, Yarasheski K, Sinha-Hikim I, Ma K, Ezzat S, Shen R, Lalani R, Asa S, Mamita M, Nair G, Arver S, Bhasin S. Organization of the human myostatin gene and expression in healthy men and HIV-infected men with muscle wasting. Proc Natl Acad Sci U S A. 1998 Dec 8;95(25):14938-43. doi: 10.1073/pnas.95.25.14938. PMID 9843994
- [Background] Schuelke M, Wagner KR, Stolz LE, Hubner C, Riebel T, Komen W, Braun T, Tobin JF, Lee SJ. Myostatin mutation associated with gross muscle hypertrophy in a child. N Engl J Med. 2004 Jun 24;350(26):2682-8. doi: 10.1056/NEJMoa040933. No abstract available. PMID 15215484
- [Background] Kazemi F. The correlation of resistance exercise-induced myostatin with insulin resistance and plasma cytokines in healthy young men. J Endocrinol Invest. 2016 Apr;39(4):383-8. doi: 10.1007/s40618-015-0373-9. Epub 2015 Aug 18. PMID 26280319
- [Background] Raue U, Slivka D, Jemiolo B, Hollon C, Trappe S. Myogenic gene expression at rest and after a bout of resistance exercise in young (18-30 yr) and old (80-89 yr) women. J Appl Physiol (1985). 2006 Jul;101(1):53-9. doi: 10.1152/japplphysiol.01616.2005. Epub 2006 Apr 6. PMID 16601301
- [Background] Kawada S, Ishii N. Skeletal muscle hypertrophy after chronic restriction of venous blood flow in rats. Med Sci Sports Exerc. 2005 Jul;37(7):1144-50. doi: 10.1249/01.mss.0000170097.59514.bb. PMID 16015131
- [Background] Brandan E, Fuentes ME, Andrade W. The proteoglycan decorin is synthesized and secreted by differentiated myotubes. Eur J Cell Biol. 1991 Aug;55(2):209-16. PMID 1935986
- [Background] Kanzleiter T, Rath M, Gorgens SW, Jensen J, Tangen DS, Kolnes AJ, Kolnes KJ, Lee S, Eckel J, Schurmann A, Eckardt K. The myokine decorin is regulated by contraction and involved in muscle hypertrophy. Biochem Biophys Res Commun. 2014 Jul 25;450(2):1089-94. doi: 10.1016/j.bbrc.2014.06.123. Epub 2014 Jul 1. PMID 24996176
- [Background] Liu MQ, Chen Z, Chen LX. Endoplasmic reticulum stress: a novel mechanism and therapeutic target for cardiovascular diseases. Acta Pharmacol Sin. 2016 Apr;37(4):425-43. doi: 10.1038/aps.2015.145. Epub 2016 Feb 1. PMID 26838072
- [Background] Guiraud S, van Wittenberghe L, Georger C, Scherman D, Kichler A. Identification of decorin derived peptides with a zinc dependent anti-myostatin activity. Neuromuscul Disord. 2012 Dec;22(12):1057-68. doi: 10.1016/j.nmd.2012.07.002. Epub 2012 Jul 31. PMID 22854012
- [Background] Bugera EM, Duhamel TA, Peeler JD, Cornish SM. The systemic myokine response of decorin, interleukin-6 (IL-6) and interleukin-15 (IL-15) to an acute bout of blood flow restricted exercise. Eur J Appl Physiol. 2018 Dec;118(12):2679-2686. doi: 10.1007/s00421-018-3995-8. Epub 2018 Sep 22. PMID 30244288

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT05573321/Prot_SAP_000.pdf